CLINICAL TRIAL: NCT06076798
Title: Clinical Performance of the AFGen1 Device Over a 7-day Period
Brief Title: Clinical Performance of AFGen1
Status: Completed | Type: Observational
Sponsor: TriVirum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 130-0006P
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Afib; ECG
Keywords: ECG signal quality
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Wear AFGen1: Wear AFGen1 for 7 days. ECG co-measurement with 12 lead device at start and end of wear period
  Interventions: Device: ECG co-measurement

INTERVENTIONS:
Device: ECG co-measurement — Measure ECG with 12 lead device at same time that AFGen1 is monitoring ECG

SUMMARY:
AFGen1 is indicated for use on symptomatic or asymptomatic adults who are at risk of developing or who have atrial fibrillation, where a software assisted analysis of ambulatory ECG is needed to identify episodes of Afib. The purpose of this study is to establish the clinical performance of AFGen1 on human participants.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate the ECG signal acquired by the AFGen1 device is of adequate quality and is suitable to support its intended use for the detection of Afib. This will be evaluated by comparing the ECG data acquired by AFGen1 to that acquired by an FDA cleared 12-lead ECG device. The study will also seek to demonstrate that there is no degradation in the quality of the ECG signal it acquires over the maximum 7-day wear period that it can be prescribed for use.

The secondary purpose of this study is to confirm the adhesive performance of the device is appropriate to support its intended use per the requirements of sections 4.4 and 5.4 of ANSI AAMI EC12-1 .

ELIGIBILITY:
Inclusion Criteria:

1. 18+ willing to sign the consent form

Exclusion Criteria:

1. Implanted pacemakers
2. Implanted cardioverter defibrillators
3. Implanted cardiac resynchronization devices
4. Potential life-threatening arrythmias
5. Physical or mental health conditions that would prevent the person from being able to follow instructions regarding participation in the study
6. Open wounds, abraded or irritated skin at the application site
7. Planned to undergo a MRI during the course of the study duration
8. Known or suspected to be pregnant
9. Student or employee of TriVirum

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study shall involve 15 participants (approximately equal number of males and females, meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Quantitative Evaluation | 7 days
  For the quantitative evaluation of the mean and standard deviation of the QRS amplitude, duration, and timing correlations for all study subjects and for the end of the wear period for those relevant subjects, the mean correlation coefficient must be greater than 0.95 and standard deviation must be less than 0.05 to validate a 95% confidence interval with significant factor of assurance.
  validate a 95% confidence interval with significant factor of assurance.
Adhesive performance | 7 days
  For the adhesive performance element of the study, the overall average wear time for the device must be greater than 5-days.

CONTACTS AND LOCATIONS:
Locations (1):
- 4927 Lillian Street, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No